CLINICAL TRIAL: NCT06421363
Title: Continuity of Care Between Primary Care Cardiology and Specialty Services for Patients With Chronic Ischemic Heart Disease
Acronym: CAPRICI
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jose Seijas Amigo (Other)
Responsible Party: Sponsor-Investigator, Jose Seijas Amigo, PhD MS Pharmacy. Head of Clinical Trial Unit of Cardiology, Hospital Clinico Universitario de Santiago
Organization: Hospital Clinico Universitario de Santiago (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CORONARIA 1/2023
Record Dates: First submitted 2024-04-24; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Ischemic Heart Disease; Acute Coronary Syndrome
Keywords: inclisiran
MeSH Terms: conditions — Myocardial Ischemia; Acute Coronary Syndrome | interventions — ALN-PCS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL GROUP (No Intervention)
- INTERVENTIONAL GROUP (Experimental)
  Interventions: Drug: Inclisiran

INTERVENTIONS:
Drug: Inclisiran — Implementation of a follow-up program that incorporates Inclisiran treatment in patients with a history of chronic coronary syndrome
  Arms: INTERVENTIONAL GROUP

SUMMARY:
1.1. Background Cardiovascular disease (CVD) remains the leading cause of death in our country for over four decades. The pathophysiology of CVD begins with various cardiovascular risk factors (CRFs) and their poor management, leading to subclinical lesions in target organs such as albuminuria or left ventricular hypertrophy, which may evolve into CVD. This progression is referred to as the cardiovascular continuum. Patients with chronic cardiovascular conditions require comprehensive periodic health monitoring in primary care (PC), including lifestyle advice and an assessment of comorbidities. Risk factors linked to disease progression are monitored and managed, along with medication reconciliation and planning follow-up care. Such activities, especially post-COVID, help maintain clinical stability and organize healthcare demand, reducing unnecessary interventions and costs. In Galicia, continuity of care programs for ischemic heart disease focus on optimizing service delivery at appropriate levels, including electronic consultations that improve healthcare accessibility, outcomes, and cost-effectiveness. Introducing Inclisiran for chronic CVD patients post-acute coronary syndrome (ACS) hospitalization might streamline care continuity, reducing healthcare costs and improving outcomes.

1.2. Purpose The disruption of care continuity in patients post-ACS increases their risk of mortality and hospitalizations due to coronary complications and comorbidities, as well as emergency visits and unplanned healthcare interactions, thus elevating healthcare costs. We propose reorganizing care continuity for ACS patients by establishing a PC pathway with scheduled semi-annual visits to assess overall and cardiovascular health and to evaluate patient prognosis and healthcare resource utilization.

2. Objectives 2.1. Primary Objectives The main goal is to evaluate whether a follow-up program incorporating Inclisiran treatment in patients with chronic coronary syndrome can optimize follow-up (reducing unscheduled visits to PC and hospital emergency departments), improve control of risk factors (like physical activity, adherence to a Mediterranean diet, lipid profiles, blood pressure, glycemic profile, and renal function), and decrease direct economic costs.

2.2. Secondary Objectives The secondary objectives include analyzing adherence to prescribed chronic pharmacological treatment, factors driving higher demand among patients with chronic coronary syndrome, reasons for emergency visits, hospital admissions, and causes of mortality among these patients.

3. Methodology 3.1. Study Design A pilot, multicentric, analytical intervention study will be conducted involving five health centers in the Santiago de Compostela health area, with specific inclusion and exclusion criteria outlined. The study will monitor patients over 27 months, following a detailed protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Prior diagnosis of chronic coronary disease

   At least one of the following:
   1. Type 2 diabetes mellitus
   2. Familial hypercholesterolemia
   3. Recurrent coronary disease
   4. Chronic kidney disease
3. Currently undergoing pharmacological treatment with high-potency statins, with or without ezetimibe. The allowed statins and daily doses are:

   1. Atorvastatin 80mg
   2. Rosuvastatin 20mg
   3. Rosuvastatin 40mg
   4. Patients on other statins or lower doses are acceptable if there has been documented intolerance to the specified molecules and doses.
4. Blood analysis with a lipid profile in the last 6 months and with the current treatment showing LDL levels >100mg/dl.

Exclusion Criteria:

1. Not receiving statins in the therapeutic regimen.
2. Concomitant treatment with PCSK9 inhibitors.
3. Pregnancy, breastfeeding, or a desire to conceive by the patient.
4. Patients who, in the opinion of the investigator, are unable to adequately follow up in the chronic care program under routine clinical practice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in Unplanned Medical Visits | 2 YEARS
  Number of unplanned visits for patients with chronic coronary syndrome in family medicine, nursing, telemedicine, and hospital consultations during follow-up.
Variation in Adherence to the Mediterranean Diet | 2 YEARS
  Change in adherence to the Mediterranean diet using the validated questionnaire PREDIMED. The test consists of 14 questions, in which the higher the score, the better the relationship with a healthy life.
  TOTAL SCORE: < 9 low adherence >= 9 good adherence to the Mediterranean diet
Change in Lipid Profile. | 2 YEARS
  Change in LDL cholesterol levels in mg/dL from baseline to follow-up. Unit of Measure: mg/dL
Change in Blood Pressure | 2 YEARS
  Change in systolic/diastolic blood pressure (specify how it's measured, e.g., mmHg).
  Unit of Measure: mmHg.

SECONDARY OUTCOMES:
Adherence to Medication | 2 YEARS
  Adherence to medication, measured as the proportion of days covered (PDC) based on the total number of days medications were supplied through the electronic prescription system.
  Unit of Measure: Percentage (%) Calculation of the PDC for a specific drug: The numerator represents the total number of days a drug was supplied between the first and last electronic prescription picked up (a + b + c + d). The denominator represents the total number of days in the interval (from x to t). PDC: proportion of days covered.
Emergency Room Attendances | 2 YEARS
  Outcome Measure: Number of hospital emergency attendances during the study period.
  Unit of Measure: Number of attendances.
Patient Prognosis | 2 YEARS
  Hospital Admissions Description: Number of hospital admissions related to cardiovascular disease Unit of Measure: Number of admissions Mortality Description: Number of deaths and primary cause during the study period. Unit of Measure: Number of admissions
Change in Patient Risk Factors | 2 YEARS
  Physical Activity Description: Change in physical activity, assessed via a validated questionnaire SF-36 Unit of Measure: Score on the questionnaire.
  Scale Details:
  Full Scale Name: Short Form (36) Health Survey Scale Range: The SF-36 scale typically ranges from 0 to 100. Interpretation: Higher scores indicate a better quality of life and health status.
Cost Analysis | 2 YEARS
  Costs associated with unplanned medical visits, adherence, hospitalizations, and medication adherence.
  Unit of Measure: Cost (currency)
Healthcare Organization 1 | 2 years
  Outcome Measure: Number of unplanned nursing consultations in primary care.
  Unit of Measure: Number of consultations.
Healthcare Organization 2 | 2 yeras
  Outcome Measure: Number of unplanned family doctor consultations in primary care.
  Unit of Measure: Number of consultations.
Healthcare Organization 3 | 2 years
  Outcome Measure: Number of attendances at continuous care points in primary care.
  Unit of Measure: Number of attendances.
Healthcare Organization 4 | 2 yeras
  Outcome Measure: Number of telemedicine hospital consultations.
  Unit of Measure: Number of consultations.
Healthcare Organization 5 | 2 years
  Outcome Measure: Number of in-person hospital consultations.
  Unit of Measure: Number of consultations.
Healthcare Organization 5 | 2 years
  Outcome Measure: Number of hospital emergency attendances.
  Unit of Measure: Number of attendances.
Lab samples results | 2 years
  Outcome Measure: Lab samples results.
  Unit of Measure: Specific measure (e.g., mg/dL for cholesterol).

CONTACTS AND LOCATIONS:
Locations (6):
- Spain (6):
  - Cenro de Salud de La Estrada, A Estrada, A Coruña
  - Centro de Salud de Milladoiro, Ames, A Coruña
  - Centro de Salud de Ribeira, Ribeira, A Coruña
  - Hospital Clinico Univesitario de Santiago de Compostela, Santiago de Compostela, A Coruña
  - Centro de Salud de Melide, Melide
  - Centro de Salud A Cañiza, Pontevedra

IPD SHARING:
Plan to Share IPD: No